CLINICAL TRIAL: NCT03826797
Title: Correlation Between Trans Esophageal Pressure and Non-invasive Respiratory Support Failure in Patients With Acute Hypoxic Respiratory Failure
Acronym: TEMPO
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 266/16; 266/16 (Other: Local Ethics Committee of Modena (Italy))
Record Dates: First submitted 2019-01-28; First posted 2019-02-01 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Failure
Keywords: Non invasive ventilation; Esophageal pressure; Transpulmonary pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at assessing the correlation between trans esophageal pressure and related respiratory mechanics (including, among others, nasal pressure-Pnose) and non-invasive respiratory support failure in patients with acute hypoxic respiratory failure of different etiology (including COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Acute hypoxic respiratory failure (P/F < 200)

Exclusion Criteria:

* Acute pulmonary edema
* Chest wall deformities
* Immediate need for Mechanical Ventilation
* Pregnancy
* Hypercapnic RF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-10-16 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Esophageal pressure impact on non invasive respiratory support (NRS) failure | 24 hours
  Correlation between esophageal pressure values within 24 hours from NRS start and NRS failure

SECONDARY OUTCOMES:
Transpulmonary pressure impact on NRS failure | 24 hours
  Correlation between transpulmonary pressure values within 24 hours from NRS start and NRS failure
Dynamic compliance impact on NRS failure | 24 hours
  Correlation between dynamic compliance values within 24 hours from NRS start and NRS failure
Dynamic mechanical power impact on NRS failure | 24 hours
  Correlation between dynamic mechanical power within 24 hours from NRS start and NRS failure
Correlation between nasal pressure (Pnose) and esophageal pressure | 24 hours
  Correlation between nasal pressure (Pnose) and esophageal pressure
Pnose impact on NRS failure | 24 hours
  Correlation between Pnose within 24 hours from NRS start and NRS failure

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Modena Policlinico, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tonelli R, Cortegiani A, Marchioni A, Fantini R, Tabbi L, Castaniere I, Biagioni E, Busani S, Nani C, Cerbone C, Vermi M, Gozzi F, Bruzzi G, Manicardi L, Pellegrino MR, Beghe B, Girardis M, Pelosi P, Gregoretti C, Ball L, Clini E. Nasal pressure swings as the measure of inspiratory effort in spontaneously breathing patients with de novo acute respiratory failure. Crit Care. 2022 Mar 24;26(1):70. doi: 10.1186/s13054-022-03938-w. PMID 35331323
- [Derived] Tonelli R, Fantini R, Tabbi L, Castaniere I, Pisani L, Pellegrino MR, Della Casa G, D'Amico R, Girardis M, Nava S, Clini EM, Marchioni A. Early Inspiratory Effort Assessment by Esophageal Manometry Predicts Noninvasive Ventilation Outcome in De Novo Respiratory Failure. A Pilot Study. Am J Respir Crit Care Med. 2020 Aug 15;202(4):558-567. doi: 10.1164/rccm.201912-2512OC. PMID 32325004